CLINICAL TRIAL: NCT06236269
Title: Prospective Biomarker Analysis in HR+/HER2- Advanced or Metastatic Breast Cancer Patients Treated With Sacituzumab Govitecan
Brief Title: HR+/HER2- Advanced or Metastatic Breast Cancer Patients Treated With Sacituzumab Govitecan
Acronym: ACROSS-TROP2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: SOLTI Breast Cancer Research Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SOLTI-2201
Record Dates: First submitted 2023-12-22; First posted 2024-02-01 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer Stage IV
Keywords: sacituzumab govitecan; breast cancer; CelTIL
MeSH Terms: conditions — Breast Neoplasms | interventions — sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sacituzumab Govitecan (Experimental): Sacituzumab govitecan will be given on Days 1, 8 of a 21-day cycle at a dose of 10 mg/kg intravenously, continuously until progression of the disease or unacceptable toxicity.
  Interventions: Drug: Sacituzumab Govitecan

INTERVENTIONS:
Drug: Sacituzumab Govitecan — Sacituzumab Govitecan 10 mg/kg will be administrad intravenously (IV) on Days 1, 8 of a 21-day cycle
  Other Names: Trodelvy

SUMMARY:
This is an open-label, single arm, non-randomized, multicenter phase II study for the identification of predictive biomarkers of sacituzumab govitecan benefit and the understanding of key resistance mechanisms in HR+/HER2- advanced/metastatic breast cancer patients

DETAILED DESCRIPTION:
This study will include patients with HR+/HER2- advanced/metastatic breast cancer who have progressed on prior endocrine therapy and CDK4/6i and who have received up to 1 prior regimen of chemotherapy or ADC for metastatic breast canncer.

The primary objective is to evaluate the change in the CelTIL score, a combined biomarker based on stromal tumor-infiltrating lymphocytes and tumor cellularity, as surrogate of treatment response after one dose of sacituzumab govitecan (SG).

Patients who fulfil all eligibility criteria will start SG at 10 mg/kg as an IV infusion on Days 1 and 8 of a 21-day cycle. SG will be administered continuously until progression of the disease, unacceptable toxicity, investigator's decision, withdrawal of consent, or other reasons described in the protocol.

Tumor tissue (newly obtained) will be sent to a central laboratory. After 2 weeks(14-21 days) of treatment a new biopsy of the same lesion will be performed. Tumor biopsy will be also performed at disease progression / EoT. In addition, blood samples (for ctDNA) will be collected at C1D1, C2D1 and at progression / EoT for exploratory objectives.

Imaging will be performed prior to day 1 of treatment and target and non-target lesions will be identified as per RECIST 1.1. Tumor assessments will be performed every 9 weeks until the start of a new anti-cancer therapy, withdrawal of consent, progression of disease, death, or the end of the study, whichever occurs first. Tumor assessments will be performed on the specified schedule regardless of treatment delays. Tumor response will be assessed as per RECIST v.1.1.

Safety assessments will include the incidence, nature, and severity of AEs and laboratory abnormalities graded per the NCI CTCAE v.5.0. Laboratory safety assessments will include the regular monitoring of hematology, blood chemistry and pregnancy test.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent form prior to any mandatory study specific procedures, sampling, and analyses.
2. Patients must be male or female (pre/peri or postmenopausal) ≥ 18 years of age.
3. ECOG performance status of 0 or 1(see Appendix 1).
4. Histologically or cytologically confirmed breast cancer with evidence of locally advanced disease, not amenable to resection or radiation therapy with curative intent or metastatic disease.
5. HR+/HER2- BC by local testing, not amenable to surgical therapy will be enrolled in this study.

   1. HER2 negativity is defined as either of the following by local laboratory assessment: IHC 0, IHC 1+ or IHC2+/in situ hybridization (ISH) negative as per the most recent American Society of Clinical Oncology (ASCO)-College of American Pathologists Guideline (CAP) guideline. If a patient has had multiple HER2 results after metastatic disease, the most recent test result prior screening period will be used to confirm eligibility.
   2. ER and/or PR positivity are defined as >1% of cells expressing HR via IHC analysis as per most recent ASCO-CAP guideline. If a patient has had multiple ER/PgR results after metastatic disease, the most recent test result prior screening period will be used to confirm eligibility.
6. Disease refractory to CDK4/6 inhibitors, defined as recurrence during or within 12 months after the end of adjuvant treatment or progression during or within 6 months after the end of treatment for advanced/metastatic disease.
7. No more than 1 prior systemic chemotherapy or antibody-drug conjugate (ADC) regimens for metastatic disease. Adjuvant or neoadjuvant therapy for early-stage disease will qualify as one of the required prior chemotherapy regimens if the development of unresectable, locally advanced, or metastatic disease occurred within a 12-month period of time of the therapy. Note: treatments for bone metastases (eg, bisphosphonates, denosumab, etc.), targeted therapies (eg, PARP inhibitors, CDK 4/6 inhibitors, immunotherapy etc.) and hormonal therapy are not considered as prior systemic chemotherapy treatments for advanced disease.
8. Radiologic or objective evidence of disease progression on or after the last systemic therapy prior to starting study treatment
9. Measurable or non-measurable disease but evaluable (identification of target and/or non-target lesions by RECIST Vs1.1).
10. Patients must have a site of disease amenable to safely perform a biopsy, as per Investigator's assessment, and be a candidate for tumor biopsy according to the treating institution's guidelines.
11. Possibility of performing a biopsy prior to the start of treatment and its repetition after 2 weeks (14-21 days) and at End of Treatment (EOT) on the same location. It will be provided formalin-fixed paraffin-embedded (FFPE) tumor block. The tumor tissue should be of good quality based on total and viable tumor content and must be evaluated centrally for quality prior to enrollment. Patients whose tumor tissue is not evaluable for central testing are not eligible. It is recommended to send the biopsy directly to the central lab after confirming the existence of a tumor, so as not to delay the inclusion, without the need to carry out IHC studies in the same sample.

    * Acceptable samples include core needle biopsies for deep tumor tissue or excisional, incisional, punch, or forceps biopsies for cutaneous, subcutaneous, bone or mucosal lesions or biopsies from bone metastases. Lymph node biopsies are also permitted.
    * Fine needle aspiration, brushing, cell pellet from pleural effusion and lavage samples are not acceptable.
12. Patients must have normal organ and bone marrow function measured within 35 days prior to administration of study treatment as defined below:

    * Haemoglobin ≥ 9.0 g/dL *
    * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L*
    * Platelet count ≥ 100 x 109/L*
    * Total bilirubin (TBL) ≤ 1.5 × upper limit of normal (ULN) or ≤ 3 × ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinemia).
    * AST (SGOT) / ALT (SGPT) ≤ 2.5 x ULN unless liver metastases are present in which case, they must be ≤ 5x ULN
    * Creatinine ≤ 1.5 x ULN or Creatinine clearance estimated of ≥30mL/min using the Cockcroft-Gault equation.
    * Serum albumin >3 g/dL
    * International normalized ratio (INR) or prothrombin time (PT) and either partial thromboplastin or activated partial thromboplastin time (aPTT) ≤ 1.5 ×ULN *Without transfusional or growth factor support within 1 week of study treatment initiation.
13. Patients must have a life expectancy ≥ 16 weeks.
14. Male patients and female patients of childbearing potential who engage in heterosexual intercourse must agree to use protocol-specified method(s) of contraception as described in Appendix 2.
15. Willing and able to comply with the requirements and restrictions in this protocol.

Exclusion Criteria:

1. Patients with HER2-positive or TNBC disease.
2. Other malignancy unless curatively treated with no evidence of disease for ≥3 years except: non-melanoma skin cancer, in situ cancer of the cervix, ductal carcinoma in situ (DCIS), Stage 1, grade 1 endometrial carcinoma or other malignant tumors with an expected curative outcome after medical monitor approval.
3. Has unresolved toxicities from previous anticancer therapy (≥ CTCAE version 5.0 grade 1) caused by previous cancer therapy, excluding alopecia or other toxicities not considered a safety risk for the patient at investigator's discretion. Note: Subjects may be enrolled with chronic, stable Grade 2 toxicities (defined as no worsening to ≥Grade 2 for at least 2 months prior to enrollment and managed with standard of care treatment) that the investigator deems related to previous anticancer therapy, such as: Chemotherapy-induced neuropathy, Fatigue, Residual toxicities from prior IO treatment Grade 1 or Grade 2 endocrinopathies. Note: if patients received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
4. Patients may not be participating in a study with an investigational agent or investigational device within 2 weeks or 5 half-lives, whichever is longer, prior to allocation. Patients participating in observational studies are eligible.
5. Patients with symptomatic uncontrolled brain metastases. Participants with a history of treated Central Nervous System (CNS) metastases are eligible, provided they meet all of the following criteria:

   * Biopsiable disease outside the CNS is present.
   * No evidence of interim CNS progression between the completion of CNS directed therapy and the screening radiographic study.
   * Metastases are limited solely to cerebellar and supratentorial lesions.
   * Stable requirement for corticosteroids (≤ 20 mg oral prednisone or equivalent) or anticonvulsants during >4 weeks as therapy for CNS disease.
   * No stereotactic radiation within 7 days or whole-brain radiation within 14 days prior to enrolment.
   * No evidence of progression or haemorrhage after completion of CNS directed therapy.
   * Patients with spinal cord compression are excluded unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days.
6. History of significant cardiovascular disease, defined as:

   * New York Heart Association Class III or greater congestive heart failure or known left ventricular ejection fraction of < 40%.
   * Unstable angina or myocardial infarction within 6 months before enrolment.
   * History of serious ventricular arrhythmia (ie, ventricular tachycardia or ventricular fibrillation), high-grade atrioventricular block, or other cardiac arrhythmias requiring antiarrhythmic medications (except for atrial fibrillation that is well controlled with antiarrhythmic medication); history of QT interval prolongation.
7. Have active chronic inflammatory bowel disease (ulcerative colitis, Crohn's disease) or GI perforation within 6 months of enrollment.
8. Have active serious infection requiring requiring IV antibiotics, antivirals, or antifungals.
9. Have a known history of Human Immunodeficiency Virus (HIV).
10. Have active HBV (defined as having a positive HbsAg test) or HCV.

    1. For patients with a history of HBV infection, a hepatitis B core antibody test should be conducted at screening. If positive, hepatitis B DNA testing will be performed and if active HBV infection is ruled out, the patient may be eligible.
    2. Patients who are HCV antibody positive with polymerase chain reaction negative for HCV RNA may be eligible.
11. Have other concurrent medical or psychiatric conditions that, in the investigator's opinion, may be likely to confound study interpretation or prevent completion of study procedures and follow-up examinations.
12. Has received a live vaccine within 30 days prior to randomization.
13. Prior treatment with Sacituzumab-govitecan.
14. Known or severe (≥ Grade 3) hypersensitivity or allergy to sacituzumab govitecan, their metabolites, or formulation excipient.
15. Requirement for ongoing therapy with or prior use of any prohibited medications listed in Section 7.5.
16. Positive serum pregnancy test or women who are lactating (see Appendix 2).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2027-02-20 (Estimated)

PRIMARY OUTCOMES:
CelTIL score | baseline and at Cycle 2 Day 1 (14-21 days after treatment initiation)
  Mean change in CelTIL score per central assessment between paired tumor samples in the overall population.
  CelTIL score = -0.8 x tumor cellularity (%) + 1.3 x tumor-infiltrating lymphocytes (TILs) (%).
  The minimum and maximum unscaled CelTIL scores will be -80 and 130. This unscaled CelTIL score will then be scaled to reflect a range from 0 to 100 points.

SECONDARY OUTCOMES:
Overall Response rate (ORR) | Until objective tumor response, assessed up to approximately 9 months
  proportion of patients with measurable disease with best overall response of complete response (CR) or partial response (PR), as per local investigator´s assessment and according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria.
Clinical Benefit Rate (CBR) | Until objective tumor response, assessed up to approximately 9 months
  Proportion of patients with a best overall response of CR, PR or an overall lesion response of Stable Disease (SD) or Non- PR/Non-progression disease (PD) lasting ≥24 weeks, based on local investigator´s assessment according to RECIST v1.1.
Progression free survival (PFS) | From date of enrollment to disease progression or death from any cause,whichever came first, assessed up to approximately 9 months
  Time from enrollment to the first occurrence of disease progression, as determined locally by the investigator through the use of RECIST v.1.1, or death from any cause, whichever occurs first.
Duration of response (DoR) | From date of enrollment to disease progression or death from any cause,whichever came first, assessed up to approximately 9 months
  Time from the first occurrence of a documented objective response to disease progression, as determined locally by the investigator through use of RECIST v.1.1, or death from any cause, whichever occurs first.
Time to response (TtR) | Until objective tumor response, assessed up to approximately 9 months
  Time from enrollment to the first objective tumor response (tumor shrinkage of ≥30%) observed for patients who achieved a CR or PR.
Correlation between baseline TROP2 expression and the variation of CelTIL score | Baseline and at the start of Cycle 2 (Day 1, cycle of 21 days)
  Correlation between TROP2 mRNA baseline levels and changes in CelTIL score at C2D1.
Correlation between TROP2 mRNA expression with TROP2 IHC expression | Baseline
  Correlation coefficients between TROP2 mRNA and TROP2 IHC biomarkers.
Correlation between baseline TROP2 IHC expression with changes in CelTIL score | Baseline and at the start of Cycle 2 (Day 1, cycle of 21 days)
  Correlation between TROP2 IHC baseline levels and changes in CelTIL score at C2D1
Clinical benefit according to TROP2 mRNA expression & TROP2 IHC expression at baseline. | Until objective tumor response, assessed up to approximately 9 months
  Association of TROP2 mRNA expression & TROP2 IHC expression at baseline with ORR.
Clinical benefit according to TROP2 mRNA expression & TROP2 IHC expression at baseline. | Until objective tumor response, assessed up to approximately 9 months
  Association of TROP2 mRNA expression & TROP2 IHC expression at baseline with CBR.
Clinical benefit according to TROP2 mRNA expression & TROP2 IHC expression at baseline. | Until objective tumor response, assessed up to approximately 9 months
  Association of TROP2 mRNA expression & TROP2 IHC expression at baseline with PFS.
Clinical benefit according to TROP2 mRNA expression & TROP2 IHC expression at baseline. | Until objective tumor response, assessed up to approximately 9 months
  Association of TROP2 mRNA expression & TROP2 IHC expression at baseline with DoR.
Clinical benefit according to TROP2 mRNA expression & TROP2 IHC expression at baseline. | Until objective tumor response, assessed up to approximately 9 months
  Association of TROP2 mRNA expression & TROP2 IHC expression at baseline with TtR.
Correlation of CelTIL score at C2D1 with long-term outcome | Until objective tumor response, assessed up to approximately 9 months
  Correlation of CelTIL score at C2D1 with ORR, CBR, PFS, DoR, TtR
Assess safety and tolerability of Sacituzumab Govitecan | Through study completion, from date of enrollment to end of study, assessed up to approximately 29 months after the first patient enrolled
  Incidence, seriousness, treatment-related and severity (grade) of Treatment Emergent Adverse Events (TEAEs) assessed by the NCI Common Terminology for Classification of Adverse Events (CTCAE) version 5, including dose reductions, delays and treatment discontinuations.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Ciruelos, MD, Principal Investigator — Hospital 12 de Octubre, Madrid/SOLTI; Mafalda Oliveira, MD, Principal Investigator — Hospital Vall d'Hebrón/SOLTI
Locations (10):
- Spain (10):
  - ICO Badalona, Badalona, Barcelona
  - ICO Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - HU Clínico San Cecilio, Granada
  - Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Sant Joan de Reus, Reus
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clínico de Valencia, Valencia